CLINICAL TRIAL: NCT04594447
Title: A Post-market,monocentric,randomised,open-label,parallel Group,prospective Clinical Study Evaluating the Functional Outcome of the Kinematic Physica KR Total Knee Replacement System Vs the Standard Physica CR Total Knee Replacement System
Brief Title: Physica System KR Vs Physica System CR (K-20)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with enrollement
Sponsor: Limacorporate S.p.a (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-20
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Replacement
Keywords: Physica KR; Physica CR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physica KR (Other): Subject that receive Physica Kinematic Retaining total Knee replacement system
  Interventions: Device: Physica Kinematic Retaining knee replacement
- Physica CR (Other): Subject that receive Physica Cruciate Retaining total Knee replacement system
  Interventions: Device: Physica Cruciate Retaining knee replacement

INTERVENTIONS:
Device: Physica Kinematic Retaining knee replacement — modular knee prosthesis with a Kinematic Retaining (KR) mechanism and posterior cruciate ligament (PCL) preservation
  Arms: Physica KR
Device: Physica Cruciate Retaining knee replacement — modular knee prosthesis with posterior cruciate ligament (PCL) preservation
  Arms: Physica CR

SUMMARY:
Post-market, monocentric, randomised, open-label, parallel group, prospective study conducted in patients who have to perform a total knee replacement (TKR) with Physica KR or Physica CR system.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the clinical, radiographic and PROMs outcomes of Total Knee Arthroplasty (TKA) with 2 Lima TKR design: Physica KR and Physica CR (randomization 1:1) from preoperative to 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of any race requiring a total knee replacement and suitable for the use of one of the two configurations of the Physica system.
2. Age ≥ 18 years old,
3. Patients who are suffering from non-inflammatory degenerative joint disease (NIDJD): including knee osteoarthritis, post-traumatic knee arthritis, avascular necrosis; or patient who are suffering from inflammatory joint disease including rheumatoid arthritis.
4. Suitable candidates for TKR who have undamaged and functional collateral ligaments
5. Suitable candidates for TKR with Physica KR and CR who have an undamaged and functional posterior cruciate ligament.
6. Patients who understand the conditions of the study and are willing and able to comply with the prescribed rehabilitation and to perform all scheduled follow-up visits.
7. Patients who have signed the Ethics Committee/IRB approved study-specific Informed Consent Form prior to the surgery.

Exclusion Criteria:

1. Patients with severe instability of the knee joint secondary to the absence of collateral ligament integrity and/or function.
2. Patients with active or any suspected infection (on the affected knee or systemic)
3. Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy
4. Patients with significant bone loss on femoral or tibial joint side
5. Current treatment for malignant and/or life-threatening nonmalignant disorders
6. Patients with known incompatibility or allergy to the product materials, and/or metal hypersensitivity to implant materials
7. Patient with open epiphyses (immature patient with active bone growth).
8. Vascular insufficiency of lower limbs severe enough to interfere with the study evaluation
9. Patients with bone stock compromised by disease, infection or prior implantation that cannot provide adequate support and/or fixation to the prosthesis
10. Patients with systemic or metabolic disorders leading to progressive bone deterioration which may impair fixation and stability of the implant
11. Any concomitant disease and dependence that might affect the performance of the implanted prosthesis
12. Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation (e.g. primary osteoporosis with significant bone loss, haemophilic disease, septicaemia, persistent acute or chronic osteomyelitis)
13. Patients who have significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery and evaluation
14. Patients who have neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
15. Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint
16. Any psychiatric illness that would prevent comprehension of the details and nature of the study
17. Patients currently participating in any other surgical intervention studies or pain management studies
18. Female patients who are pregnant, nursing, or planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Baseline to 1 year FU
  Changes of the Oxford Knee Score (OKS) from preoperative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
  Specifically designed and developed to assess function and pain after TKR surgery. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.

SECONDARY OUTCOMES:
30-second Chair Stand Test (30 CST) | Baseline to 1 year FU
  Functional changes in 30-second Chair Stand Test (30 CST) from pre-operative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
40 metre fast paced walk test | Baseline to 1 year FU
  Functional changes in 40 metre fast paced walk test from preoperative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline to 1 year FU
  Changes in the Knee injury and Osteoarthritis Outcome Score (KOOS) from pre-operative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
  KOOS is a 42-item self-administered self-explanatory questionnaire that covers five patient-relevant dimensions: Pain, Other Disease-Specific Symptoms, Active Daily Living Function, Sport and Recreation Function, and knee-related Quality of Life. A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems
Medical Outcomes Survey Short Form-36 (SF-36) RAND SF-36 | Baseline to 1 year FU
  Changes in 36-Item Short Form Health Survey (SF-36) outcome from pre-operative (baseline) to 1 year after the implant.
  This questionnaire includes 8 scales of differing domains of health: physical functioning, bodily pain, role-physical, general health, vitality, role emotional, social functioning, and mental health. Each scale is scored on a 0 to 100 scale with a 100 representing the best score possible.
Forgotten Joint Score (FJS) | Baseline to 1 year FU
  Changes in the Forgotten Joint Score (FJS) from pre-operative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
  It comprises measures for the assessment of joint-specific patient-reported outcome and focus on patients' awareness of a specific joint in everyday life. It consists of 12 questions and is scored using a 5-point Likert response format (never-almost never-seldom- sometimes-mostly) with the raw scores transformed onto a 0-100 point scale. High scores indicate good outcome.
Range of Motion (ROM) | Baseline to 1 year FU
  Changes in the Range of Motion (ROM) from pre-operative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
Knee Society Score (KSS) | Baseline to 1 year FU
  Changes in the Knee Society Score (KSS) from pre-operative (baseline) to 1 year after the implant of the Physica KR compared to Physica CR designs.
  KSS is divided into two components to assess the knee clinically through the physical examination, and to assess the individual's functionality . The maximum score of 100 points that is the best outcome.
Radiographic evaluation | Baseline to 1 year FU
  Radiographic implant evaluation and stability assessment of the Physica KR compared to Physica CR designs at baseline and 1 year after the implant.
Serious Adverse Event (SAE) incidence | Baseline to 1 year FU
  Changes Incidence, type and severity of all device-related Serious Adverse Events (SAEs) at intra-operatively, at discharge, 6 months and 1 year after the implant.
Adverse Event (AE) device related incidence | Baseline to 1 year FU
  Incidence, type and severity of all device-related Adverse Events (AEs) at intraoperatively, at discharge, 6 months and 1 year after the implant

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No